CLINICAL TRIAL: NCT05312905
Title: Home-based Mirror Therapy and Cognitive Therapeutic Exercises After Stroke
Brief Title: Mirror Therapy in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Farzin Hajebrahimi, PhD, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MirrorCog2021
Record Dates: First submitted 2022-03-14; First posted 2022-04-06 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Cognitive Therapy; Telerehabilitation
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be included in the study and randomly divided into two groups using block randomization in Microsoft Excel-RANDOMISE 'RAND(WS)' function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Active Comparator): Exercises including mirror therapy will be applied to the participants in the Mirror Therapy group. The mirror will be placed in such a way that the affected extremity of the patient could not be seen behind the mirror and the healthy extremity would be in front of his eyes, the patient will perform the exercises indicated by the physiotherapist with his intact extremity, looking into the mirror. The exercises will be performed in sessions lasting 60 minutes, 3 days a week, over 8 weeks.
  Interventions: Other: Mirror Therapy
- Mirror+Cognitive Therapy (Experimental): The participants in the Mirror+Cognitive Therapy will be given a cognitive task with the application of mirror therapy. Cognitive tasks with mirror therapy will be applied in sessions lasting 60 minutes, 3 days a week, over 8 weeks.
  Interventions: Other: Mirror Therapy + Cognitive Therapy

INTERVENTIONS:
Other: Mirror Therapy — Mirror Therapy applied alone
  Arms: Mirror Therapy
Other: Mirror Therapy + Cognitive Therapy — Mirror Therapy supported with Cognitive Exercises
  Arms: Mirror+Cognitive Therapy

SUMMARY:
Little is known about mirror therapy and cognitive exercises applied together in patients with stroke by means of telerehabilitation. The aim of this study is to investigate the effects of home-based mirror therapy combined with cognitive exercises on upper extremity functions and cognition in adults with stroke and to compare these effects with mirror therapy alone.

ELIGIBILITY:
Inclusion Criteria:

Age 40 years old and over having had a stroke having unilateral involvement having sufficient communication skills to answer oral and written questions and following instructions 20< points in MMSE

Exclusion Criteria:

a stroke history under the age of 40 not having a verbal or written communication level that cannot fulfill the study conditions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | changes after 8 weeks
  The Mini-Mental State Examination (MMSE) is a 30-point test. Higher values mean better performance.
Fugl-Meyer Upper Extremity Motor Assessment | changes after 8 weeks
  The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. The total possible scale score is 226. Higher scores mean better performance.

SECONDARY OUTCOMES:
Stroke-Specific Quality of Life Scale | changes after 8 weeks
  Specific Quality Of Life scale (SSQOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. The original test consists of 49 items encompassing 12 domains. Each item is ranked on a 5-point scale, with higher scores indicating better function.
Beck Depression Scale | changes after 8 weeks
  The Beck Depression Scale is a 21-item self-report inventory designed to assess the presence and severity in depressive symptoms. Each item is rated on a 4-point Likert-type scale ranging from 0 to 3, based on the severity in the last two weeks. Higher scores indicating worse level of depression.
Barthel Activity of Daily Living Scale | changes after 8 weeks
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Eight factors are rated to produce an overall score on a point scale of 0 to 100. Then, an assignment is given as "excellent" for 95 to 100 points; "good" for 84 to 94 points, "fair" for 65 to 83 points, or "poor" for less than 65 points, higher scores indicating better function.
Modified Ashworth Scale | changes after 8 weeks
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform.This scale grades the muscle tone from 0 (normal) to 4 (severe spasticity). The usage of this scale is easy; however, the results depend on the evaluator. Higher scores indicating sever spasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on reasonable request from the Principle Investigator. The data are not publicly available due to ethical issues.